CLINICAL TRIAL: NCT03455140
Title: A Phase I/II Study Evaluating the Safety and Activity of Pegylated Recombinant Human Arginase (BCT-100) in Relapsed/Refractory Cancers of Children and Young Adults
Brief Title: A Study Evaluating the Safety and Activity of Pegylated Recombinant Human Arginase (BCT-100)
Acronym: PARC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG_16-040
Record Dates: First submitted 2018-02-01; First posted 2018-03-06 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Cancer; Pediatric Solid Tumor; Pediatric AML; Pediatric ALL
Keywords: Arginine; Arginase; Children; Young Adult
MeSH Terms: conditions — Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — BCT-100

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 - Leukaemia (Experimental): PEG- BCT-100 in patients with Leukaemia Starting dose 1600U/Kg IV infusion weekly
  Interventions: Drug: PEG- BCT-100
- Group 2 - Neuroblastoma (Experimental): PEG- BCT-100 in patients with Neuroblastoma Starting dose 1600U/Kg IV infusion weekly
  Interventions: Drug: PEG- BCT-100
- Group 3 - Sarcomas (Experimental): PEG- BCT-100 in patients with Sarcomas Starting dose 1600U/Kg IV infusion weekly
  Interventions: Drug: PEG- BCT-100
- Group 4 - High Grade Glioma (Experimental): PEG- BCT-100 in patients with High Grade Gliomas Starting dose 1600U/Kg IV infusion weekly
  Interventions: Drug: PEG- BCT-100

INTERVENTIONS:
Drug: PEG- BCT-100 — PEGylated recombinant human arginase 1
  Other Names: rhArg1peg5000

SUMMARY:
PARC is an international phase I/II trial evaluating the safety and activity of pegylated recombinant human arginase (BCT-100) in children and young people with relapsed/refractory leukaemia, neuroblastoma, sarcoma and high grade gliomas (brain cancers).

Currently the outcomes for these patients are poor and the therapeutic options are limited with a significant toxicity burden. Therefore new treatments which work in different ways to standard chemotherapy are urgently needed. Research has shown that arginine (a nutrient) is important in the survival of cancer cells. BCT-100 is a drug which can deplete arginine levels and starve cancer cells - a completely new approach. BCT-100 has been tested in adults and shown to be active with almost no side-effects. This trial will test whether this dose of BCT-100 is also safe and active in children with relapsed/refractory leukaemia, neuroblastoma, sarcoma and high grade glioma. The trial will also study how BCT-100 is broken down in the body and look for new biological markers of treatment response. Up to 64 children with relapsed cancers will be recruited over 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Aged 1- <25 years old at the time of study registration
* Histologically confirmed disease in one of the following four groups:

  * Group 1 - Acute lymphoblastic leukaemia (ALL) and acute myeloid leukaemia (AML)
  * Group 2 - Neuroblastoma Group 3 - Sarcoma
  * Group 4 - High grade glioma (as defined by 2016 WHO CNS classification)
* Radiological or laboratory evidence of disease progression (during or after completion of first line treatment) or any subsequent recurrence (biopsy at relapse is not mandated).
* Measurable bone marrow disease (group 1) or at least one evaluable radiological site of disease (group 2, 3 and 4).
* Adequate liver function defined as a total bilirubin ≤1.5x the upper limit of normal for age and ALT ≤ 3x the upper limit of normal for age
* Documented negative pregnancy test for female patients of childbearing potential within 7 days of trial entry
* Sexually active patients must agree to use adequate and appropriate contraception while on study drug and for 12 months following treatment discontinuation
* Written informed consent given by patient and/or parents/legal representative

Exclusion Criteria:

* Previous treatment with another therapeutic arginine depleting drug (bacterial or human) or arginase inhibitor
* Presence of any ≥ CTCAE grade 3 clinically significant treatment-related toxicity from prior therapies
* Pregnant or lactating female
* Evidence of uncontrolled infection

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 49 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2022-07-22 (Actual)

PRIMARY OUTCOMES:
Phase I: to establish the recommended phase II dose (RP2D) of BCT-100 in children and young adults as assessed by dose limiting toxicity (DLT) and complete arginine depletion | 28 days
  Safety profile as measured by the occurrence/non-occurrence of DLT within 28 days of treatment with BCT-100.
  o Optimal dose as measured by the complete depletion of arginine. This is defined as AAD <8μM arginine in the blood after 3 doses of BCT-100.
Phase II: to determine the activity of single agent BCT-100 against relapsed/refractory leukaemia, neuroblastoma, sarcoma and high grade glioma in children and young adults as measured by disease response after 8 weeks. | After 8 weeks
  Disease response (Complete Response (CR) or Partial Response (PR)) after 8 weeks of treatment with BCT-100

SECONDARY OUTCOMES:
The incidence and severity of Adverse Events (AEs) as Assessed by CTCAE v4 | 28 days after treatment completion
  Incidence and severity of Adverse Events (AEs) defined by National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v4
Disease response - Leukaemia | Within 1 year
  Disease response ( CR / PR) according to Cheson criteria
Disease response - Sarcoma | Within 1 year
  Disease response ( CR / PR) according to RECIST criteria
Disease response - High Grade Glioma | Within 1 year
  Disease response ( CR / PR) according to RANO criteria
Disease response - Neuroblastoma | Within 1 year
  Disease response ( CR / PR) according to INCR criteria
Progression free survival (PFS) | Up to three years after registration
Overall survival (OS). | Up to three years after registration
Maximum Plasma Concentration [Cmax], of BCT-100 in the paediatric population. | Up to 24 weeks
Time to maximum Plasma Concentration [Tmax], of BCT-100 in the paediatric population. | Up to 24 weeks
Minimum Plasma Concentration [Cmin], of BCT-100 in the paediatric population. | Up to 24 weeks
Area Under the Curve [AUC], of BCT-100 in the paediatric population. | Up to 24 weeks
Duration of adequate arginine depletion in blood. | Up to 24 weeks
  BCT-100 concentration in blood
Duration of adequate arginine depletion in bone marrow . | Up to 24 weeks
  BCT-100 concentration in bone marrow
Duration of adequate arginine depletion in cerebrospinal fluid. | Up to 24 weeks
  BCT-100 concentration in cerebrospinal fluid

CONTACTS AND LOCATIONS:
Overall Officials: Francis J Mussai, DPhil, Study Chair — University of Birmingham
Locations (14):
- Australia (6):
  - Women's & Children's Hospital, Adelaide
  - Queensland Children's Hospital, Brisbane
  - Royal Children's Hospital Melbourne, Melbourne
  - Perth Children's Hospital, Perth
  - Children's Hospital Westmead, Sydney
  - Sydney Children's Hospital, Sydney
- Princes Maxima Centrum, Utrecht, Netherlands
- United Kingdom (7):
  - Birmingham Children's Hospital, Birmingham
  - Bristol Royal Hospital for Children, Bristol
  - Addenbrookes Hospital, Cambridge
  - Royal Hospital for Children, Glasgow
  - Leeds Children's Hospital, Leeds
  - Royal Manchester Children's Hospital, Manchester
  - Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fenwick N, Weston R, Wheatley K, Hodgson J, Marshall L, Elliott M, Makin G, Ng A, Brennan B, Lowis S, Adamski J, Kilday JP, Cox R, Gattens M, Moore A, Trahair T, Ronghe M, Campbell M, Campbell H, Williams MW, Kirby M, Van Eijkelenburg N, Keely J, Scarpa U, Stavrou V, Fultang L, Booth S, Cheng P, De Santo C, Mussai F. PARC: a phase I/II study evaluating the safety and activity of pegylated recombinant human arginase BCT-100 in relapsed/refractory cancers of children and young adults. Front Oncol. 2024 Jan 31;14:1296576. doi: 10.3389/fonc.2024.1296576. eCollection 2024. PMID 38357205